CLINICAL TRIAL: NCT03549585
Title: End-of-Life Patient Identification Assistance in Acute GEriatric Medicine: Construction and Validation of a Prognostic Tool
Brief Title: End-of-Life Patient Identification Assistance in Acute GEriatric Medicine
Acronym: ARPEGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7732; 2016-A00116-45 (Other: ID-RCB)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Old Age
Keywords: End of life; Spotting; Emergency; criSTAL
MeSH Terms: conditions — Death; Metrorrhagia; Emergencies | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Criteria for Screening and Triaging to Appropriate aLternative care — CriSTAL Tool (Criteria for Screening and Treatment of Appropriate Long-Term Care) is a multidimensional geriatric tool that lists 18 elements of the literature, under construction and validation by an Australian retrospective study. This tool is a practical questionnaire and easy to use in current care, with items adapted to the geriatric dimension. The investigators chose to target hospitalized geriatric patients through emergencies.

SUMMARY:
The main objective of this project is to build a tool, adapted to the French geriatric population, that will predict the risk of death at three months after hospitalization in acute geriatric medicine. This tool will be built using selected items via a review of the literature published in 2015.

The 8 items of the CriSTAL tool will be collected prospectively in all patients hospitalized successively in the 2 post-emergency geriatric services (PUG) of the University Hospital of Toulouse, over a period of 9 months, by a dedicated clinical research associate. Patient survival will be assessed by obtaining the vital status of the cohort via CépiDC

DETAILED DESCRIPTION:
As the population ages, the prevalence of chronic diseases increases. Let's take the example of cardiovascular, respiratory or neurological diseases, including Alzheimer's disease. These pathologies are at the origin of decompensations requiring sometimes multiple hospitalizations. It is clear that the goals of care (curative or palliative) are not always related to life expectancy. Decision making, especially in an acute context, is often tricky. The use of a tool with certain parameters of the patient could help to guide the reflection. The present study propose a tool proposed by an Australian team (CriSTAL), which lists items described in the literature as a risk factor for the death of elderly patients. This tool is currently being studied in several types of populations around the world (general population, cancer patients, hospitalized etc.).

This is a prospective study aimed at evaluating routine, single-center care, conducted at Toulouse University Hospital.

The successive inclusion of hospitalized patients in Post Emergencies Geriatric (PUG) unity will be carried out over a period of 9 months.

The primary outcome will be the vital status (alive / deceased) at 3 months of hospitalization in acute geriatric medicine.

ELIGIBILITY:
Inclusion Criteria:

* Any geriatric patient hospitalized via emergencies at Post Emergencies Geriatric (PUG) unity
* Oral agreement of non-opposition to the use of the data relative to their hospitalization and relative to their evolution within 3 months following the hospitalization

Exclusion Criteria:

* Patient having expressed his opposition to the use of data related to his hospitalization

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive patients above 65 years old hospitalized in the 2 departments of PUG Toulouse of University Hospital will be included, over a period of 9 months.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The vital status (alive / deceased) at 3 months | 3 months
  The vital status (alive / deceased) at 3 months of hospitalization in acute geriatric medicine.Survival will be collected in a data base.

SECONDARY OUTCOMES:
The 8 items of the CriSTAL tool | 3 months
  Socio-demographic data of the geriatric patient in the emergencies
The 8 items of the CriSTAL tool | 3 months
  The reason for admission of geriatric patients in the emergencies
The 8 items of the CriSTAL tool | 3 months
  The variables potentially associated with the three-month death like Cognitive impairment
The 8 items of the CriSTAL tool | 3 months
  The variables potentially associated with the three-month death : Hospitalization in intensive care during the last year
The 8 items of the CriSTAL tool | 3 months
  ECG anomaly : ACFA, tachycardia, rhythm disorder> 5 per min, Q or ST segment abnormality

CONTACTS AND LOCATIONS:
Overall Officials: Fati Nourhashemi, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steinmeyer Z, Piau A, Thomazeau J, Kai SHY, Nourhashemi F. Mortality in hospitalised older patients: the WHALES short-term predictive score. BMJ Support Palliat Care. 2021 Nov 25:bmjspcare-2021-003258. doi: 10.1136/bmjspcare-2021-003258. Online ahead of print. PMID 34824134